CLINICAL TRIAL: NCT01110746
Title: A Double-blind Study of the Effect on Post-prandial Glycemia Safety, and Tolerability of Viaject 7 vs. Lispro Insulin During Subcutaneous Insulin Pump Therapy
Brief Title: To Evaluate the Effect on Post-prandial Glycemia Safety, and Tolerability of Viaject 7 vs. Lispro Insulin During Subcutaneous Insulin Pump Therapy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Biodel (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: VIAject -032J
Record Dates: First submitted 2010-04-13; First posted 2010-04-27 (Estimated); Last update posted 2015-08-03 (Estimated); Status verified 2015-07

CONDITIONS: Type 1 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Insulin Lispro

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Formulation A (Experimental): Single Injection
  Interventions: Drug: Viaject 7
- Formulation B (Experimental): Single Injection
  Interventions: Drug: LISPRO

INTERVENTIONS:
Drug: Viaject 7 — 100IU/mL administered subcutaneously
  Arms: Formulation A
Drug: LISPRO — 100IU/mL administered subcutaneously
  Arms: Formulation B

SUMMARY:
The purpose of this study is to evaluate the Effect on Post-prandial Glycemia Safety, and Tolerability of Viaject 7 vs. Lispro Insulin during SC Insulin Pump Therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females diagnosed with type 1 diabetes mellitus for at least 6 months
2. Current usage of subcutaneous insulin pump treatment with one of the following pumps:

   * Medtronic Paradigm®
   * Animas®
   * OmniPod®
   * ACCU-CHEK Spirit®
3. Age 18-75 years
4. HbA1c of 6.0 - 9.0% at screening visit.
5. Willingness to attend 9 clinic visits.

Exclusion Criteria:

1. Pregnancy or Lactation
2. Renal insufficiency (serum creatinine of 2.0 mg/dL or greater).
3. Anemia
4. Congestive heart failure.
5. Visual impairment preventing reading of glucose meter values or the ability to use an insulin pump or continuous glucose monitoring device.
6. Active coronary artery disease or heart procedure within the past 4 months.
7. Active foot ulceration.
8. Severe peripheral arterial disease.
9. Stroke within the past 6 months.
10. Active alcohol abuse, substance abuse, or severe mental illness.
11. Active cancer, except basal cell or squamous cell skin cancers.
12. Major surgical operation within 30 days prior to screening.
13. Seizure disorder (epilepsy).
14. Any concurrent illness, other than diabetes, that is not controlled by a stable therapeutic regimen.
15. Currently use of corticosteroids.
16. History of major non-compliance.
17. Use of an investigational drug within 30 days prior to screening.
18. Bleeding disorder, treatment with warfarin, or low platelet count.
19. Any insulin allergy
20. Current complaints of major infusion site problems with commercially- available insulin preparations, such as frequent occurrence of infections, marked swelling or marked erythema.
21. History of gastroparesis.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2010-02; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
3 hour incremental area under the glucose curve after a standardized high glycemic index meal. | 3 hours

SECONDARY OUTCOMES:
Draize scores at insulin infusion site at 24 hour and 72 hour follow-up visits, frequency of discomfort with insulin infusion, and severity of discomfort with insulin infusion (ratings of mild, moderate, or severe). | 72 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Oregon Health and Science University/Legacy Health System, Portland, Oregon, United States